CLINICAL TRIAL: NCT01443039
Title: Phenotypical Approach of the Drug Metabolizing Hormones Activity (CYP1A2, CYP2D6, CYP2C9, CYP2C19, CYP3A4 and P-gp) Before and After Roux-en Y-Gastric Bypass. The SODA Protocol: Surgery for Obesity and Drug Availability
Brief Title: Phenotypical Approach of the Drug Metabolizing Hormones Activity Before and After Roux-en Y-Gastric Bypass
Acronym: SODA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P100506; 2011-A00312-39 (Other: IDRCB)
Record Dates: First submitted 2011-08-19; First posted 2011-09-29 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Obesity
Keywords: drug metabolizing enzymes and drug transporter; Roux-en Y-Gastric Bypass; Obesity; Drug Availability; BMI over 35kg/m² and comorbidities or >40kg/m²
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- phenotypical approach (Experimental): phenotypical approach
  Interventions: Drug: phenotypical approach

INTERVENTIONS:
Drug: phenotypical approach — each visit : CAFEINE : (solution orale) 2 ampoules de 2 ml = 100 mg de CAFEINE DEXTROMETHORPHANE : 15 ml de sirop contains 20 mg =>22,5 ml = 30mg Midazolam : (solution injectable, ampoule 1 ml = 1 mg) : deux ampoules = 2 mg Digoxine nativelle (solution injectable, ampoule de 0.5mg) : 1 ampoule per os = 0.5 mg Losartan 50 mg : 1cp de 50mg

SUMMARY:
The activity of drug-metabolizing enzymes and transporters evolutes after Roux-en-Y gastric Bypass.

Primary aim : To study the intra individual evolution of phenotypical markers of different drug metabolizing enzymes and one transporter (CYP1A2, CYP2D6, CYP2C9, CYP2C19, CYP3A4 and P-gp), using a cocktail phenotypic approach, after Roux-en-Y gastric Bypass.

DETAILED DESCRIPTION:
Principal Judgement criteria :

Phenotypical markers of enzymes and transporter activity before, at 5-8 weeks and 25-30 weeks following surgery.

Secondary judgement criteria :

* Genetic polymorphisms known to affect expression and/or activity of enzymes and transporter.
* Intestinal and hepatic expression and activity of the enzymes and transporter of interest.
* Markers of inflammation Methodology, study design : open-labelled monocentric study.

Sample size : It will be a descriptive experimental study involving 12 subjects.

Study design : In centre 1: Inclusion at least 2 weeks prior to surgery (V0)

In centre 2: Three studies of 12 hours each will occur (in addition with the usual clinical and surgical follow up) at three times periods: in the 8 weeks period before surgery (V1), at 5-8 weeks after surgery (V2) and at 25-30 weeks after surgery (V3).

In centre 3: the patients will undergo gastric bypass surgery (corresponding to the usual clinical and surgical follow up) and samples of jejunum and liver will be obtain during the surgery (J0).

Centres 4 and 5 are involved in samples analysis.Hence, patients will attend 3 visits, in addition to the usual clinical and surgical follow-up.

Study duration: 26 months (with duration of inclusion of 18 months)

Duration for a patient: 38 weeks at maximum (8 months)

Investigating center and participating units: one center enrolling the patients and three centers involving in the others investigations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with morbid obesity (IMC > 40 kg/m²) or severe obesity (IMC=35-40 kg/m²) with co morbidities (sleep apnea syndrome or hypertension without treatment or steatosis hepatitis) candidates for a gastric bypass.
* Patient not receiving more than two treatments whose effect on the expression of enzymes and drug transporters is zero other than vitamins.
* Patient agreeing to participate at three studies of one day (12 hours) occurring at three different periods.
* Patients aged between 18 and 60 years old.
* Patient giving its well-informed and free consent.
* Patient without allergy to any of the drugs used for test.
* Patients living in France during the study and with French social security

Exclusion Criteria:

* Tabacco
* Contraception including estrogens compounds
* Medication other than vitamins.
* Allergy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2011-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Phenotypical markers of enzymes and transporter activity | at 5-8weeks
  plasmatic [Paraxanthine/caffeine] ratio (T4H) at 5-8 weeks following surgery. - plasmatic [Omeprazole/5-hydroxyomeprazole] ratio (T4H) at 5-8 weeks following surgery. - urinary Log (dextromethorphan/dextrorphan) (T0-T8h) at 5-8 weeks following surgery. - urinary Losartan/ E-3174 (T0-8h) at 5-8 weeks following surgery. - plasmatic AUC 0-inf midazolam at 5-8 weeks following surgery. - plasmatic AUC 0-inf digoxin at 5-8 weeks following surgery
Phenotypical markers of enzymes and transporter activity | 25-30 weeks
  plasmatic [Paraxanthine/caffeine] ratio (T4H) at 25-30 weeks following surgery. - plasmatic [Omeprazole/5-hydroxyomeprazole] ratio (T4H) at 25-30 weeks following surgery. - urinary Log (dextromethorphan/dextrorphan) (T0-T8h) at 25-30 weeks following surgery. - urinary Losartan/ E-3174 (T0-8h) at 25-30 weeks following surgery. - plasmatic AUC 0-inf midazolam at 25-30 weeks following surgery. - plasmatic AUC 0-inf digoxin at 25-30 weeks following surgery

SECONDARY OUTCOMES:
Intestinal and hepatic expression and activity of the enzymes and transporter of interest and markers of inflammation | before surgery
  Intestinal and hepatic expression and activity of the enzymes and transporter of interest and markers of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Célia LLORET-LINARES, MD,, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Unit of internal medicine A, Lariboisière Hospital, Paris, France